CLINICAL TRIAL: NCT06530316
Title: The Efficacy and Safety of RET Inhibitor for Neoadjuvant Therapy in Locally Advanced RET-altered Thyroid Cancer: a Real-world Study
Brief Title: RET Inhibitor for Neoadjuvant Therapy in Locally Advanced RET-altered Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Wang, Chief of Head and Neck Surgery, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: PATHYOID
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- None MTC: DTC, PDTC and ATC patients with RET fusions.
  Interventions: Drug: RET Inhibitor; Procedure: Surgery
- MTC: MTC patients with RET mutations
  Interventions: Drug: RET Inhibitor; Procedure: Surgery

INTERVENTIONS:
Drug: RET Inhibitor — RET inhibitors for neoadjuvant treatment
Procedure: Surgery — Operable patients receive surgery after neoadjuvant therapy

SUMMARY:
This study is a multicenter observational study. Patients receive neoadjuvant therapy with RET inhibitors in the real world, and those who can undergo surgery after neoadjuvant therapy receive surgical treatment. The aim of the study is to determine the efficacy and safety of RET inhibitors for neoadjuvant therapy in locally advanced RET-altered thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily join this study and sign an informed consent form;
* Age: ≥ 14 years old, male or female not limited;
* Locally advanced thyroid cancer diagnosed by histopathology, including papillary thyroid carcinoma, medullary thyroid carcinoma, follicular thyroid carcinoma, poorly differentiated/poorly differentiated thyroid carcinoma, etc;
* RET alterations, including fusion and mutations;
* The definition of locally advanced thyroid cancer meets at least one of the following criteria:

  1. Local advanced thyroid cancer with estimated surgical difficulty and inability to R0/1 resection;
  2. T4 thyroid cancer defined by AJCC: any size of tumor primary lesion or regional lymph node infiltration beyond the thyroid capsule to subcutaneous soft tissue, larynx, trachea, esophagus, or recurrent laryngeal nerve, tumor invasion of pre vertebral fascia or wrapping around carotid or mediastinal blood vessels;
  3. According to the imaging score, the resectable probability is less than 80% based on CT.
* At least one measurable lesion;
* For patients with distant metastasis, researchers need to determine whether patients would benefit from surgery;
* Patients voluntarily undergo tumor tissue biopsy/surgery during enrollment and withdrawal;
* Normal function of major organs.

Exclusion Criteria:

* Previously used RET inhibitors;
* There are multiple factors that affect the absorption of oral medication, such as inability to swallow, nausea and vomiting, chronic diarrhea, and intestinal obstruction;
* The patient refuses to undergo tumor tissue biopsy or surgery;
* Patients who are unsuitable for RET inhibitors or surgery.

Ages: 14 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally advanced thyroid cancer and RET alterations, who require RET inhibitor treatment and surgery after neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
R0/1 resection rate | 1 year

SECONDARY OUTCOMES:
Objective Response Rate, ORR | 1 year
Disease Control Rate，DCR | 1 year
Time to objective response，TTR | 1 year
Progression Free Survival，PFS | 5 years
Overall Survival，OS | 5 years
Adverse Events | During RET inhibitor treatment, up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Univeristy Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided